CLINICAL TRIAL: NCT03062475
Title: The Efficacy of Lifestyle Intervention in Preventing the the Recurrence of Gestational Diabetes Mellitus
Brief Title: Lifestyle Intervention to Prevent the Recurrence of Gestational Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Wang Chen, Principle investigator, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20170226
Record Dates: First submitted 2017-02-11; First posted 2017-02-23 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Gestational Diabetes Mellitus (GDM)
MeSH Terms: conditions — Diabetes, Gestational | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lifestyle intervention group (Experimental): Pregnant women allocated to this group receive lifestyle intervention. With the dietary intervention we aimed to promote a healthy pattern of eating but not necessarily to restrict energy intake. With respect to advice on physical activity, we focused on incremental increases in walking from a pedometer assessed or encourage them to do moderate cycling.
  Interventions: Behavioral: lifestyle intervention with dietary and exercise recommendation
- control group (No Intervention): Pregnant women allocated to this group receive standard prenatal care.

INTERVENTIONS:
Behavioral: lifestyle intervention with dietary and exercise recommendation — With the dietary intervention we aimed to promote a healthy pattern of eating but not necessarily to restrict energy intake.For example we suggested exchanging carbohydrate-rich foods with a medium-to-high glycaemic index for those with a lower glycaemic index to reduce the glycaemic load, and restricting dietary intake of saturated fat.
  With respect to advice on physical activity, we focused on incremental increases in walking from a pedometer assessed, or encourage them to do moderate cycling during pregnancy.
  Arms: lifestyle intervention group

SUMMARY:
Gestational diabetes mellitus(GDM) is a commom complication during pregnancy and associated with various adverse pregnancy outcomes for both the mother and her offspring. Imoportantly, with the gradual opening of a two-child policy, more and more Chinese women of reproductive age enter pregnancy have a history of GDM. Our previous study showed that regular exercise commenced in early pregnancy is effective in reducing the risk of developing GDM in Chinese overweight and obese pregant women. Thus, in this study, we want to evaluate the effect of lifestyle intervention with detailed information on how to eat and how to diet in preventing the recurrence of GDM.

DETAILED DESCRIPTION:
Gestational diabetes mellitus(GDM) is a commom complication during pregnancy. and the incidence has reached as high as 19.2% in China. GDM is associated with various adverse pregnancy outcomes for both the mother and her offspring, and not only during the perinatal phase, but also in the long term.Thus finding effective way to reduce the risk of GDM is of great importance,especial for women with high GDM risk factors. GDM history is one of the risk factors. Imoportantly, with the gradual opening of a two-child policy, more and more Chinese women of reproductive age enter pregnancy have a history of GDM. Our previous study showed that regular exercise commenced in early pregnancy is effective in reducing the risk of developing GDM in Chinese overweight and obese pregant women. Thus, in this study, we want to evaluate the effect of lifestyle intervention with detailed information on how to eat and how to diet in preventing the recurrence of GDM

ELIGIBILITY:
Inclusion Criteria:

* Singleton;
* non-smoking ;
* before 12+6 weeks gestation.

Exclusion Criteria:

* less than 18 years old;
* unwilling to provide informed consent;
* cervical insufficiency;
* women on any medication for pre-existing hypertension, diabetes, cardiac disease, renal disease, systemic lupus erythematosus, thyroid disease or psychosis;
* women who were currently being treated with metformin or corticosteroids.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 660 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
GDM | 24-28 gestational weeks
  According to the new criteria amended in August 2014 in China, GDM was diagnosed when any one value reaches or exceeds 5.1 mmol/L at 0 hours, 10.0 mmol/L at 1 hour, or 8.5 mmol/L at 2 hours. Values of 7.0 mmol/L at 0 hours or 11.1 mmol/L at 2 hours were diagnosed as DM, regardless of the pregnancy stage

SECONDARY OUTCOMES:
birth weight | up to 43 gestational weeks
  birth weight measured after baby was delivered and accurate to 0.1 kg
gestational weeks | up to 43 gestational weeks
  record the gestational weeks for delivery
delivery mode | up to 43 gestational weeks
  this includes vaginal delivery, operative vaginal delivery or cesarean delivery
macrosomia | up to 43 gestational weeks
  birth weight above 4000.0 g
LGA | up to 43 gestational weeks
  birth weight above the 90th percentile for gestational age
SGA | up to 43 gestational weeks
  birth weight below the 10th percentile for gestational age
gestational hypertention | up to 43 gestational weeks
  defined as blood pressure elevation [systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg] after 20 weeks gestation in the absence of proteinuria
pre-eclampsia | up to 43 gestational weeks
  defined as new-onset hypertension [systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg] and new-onset proteinuria [300 mg of protein in 24 hours or a urine protein/creatinine ratio of 0.3 mg/dL] after 20 weeks gestation or, in the absence of proteinuria, new-onset hypertension with new-onset thrombocytopenia, renal insufficiency, impaired liver function, pulmonary edema, or cerebral or visual disturbances

CONTACTS AND LOCATIONS:
Overall Officials: Huixia Yang, Study Chair — Peking Unviersity First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided